CLINICAL TRIAL: NCT06512532
Title: Fireworks Eye Injuries During Festivals in Upper Egypt: Cross- Sectional Study
Brief Title: Fireworks Eye Injuries During Festivals in Upper Egypt
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma Mohamed M. A. Kedwany, associate professor, Assiut University
Other Study IDs: Firework eye injury
Record Dates: First submitted 2024-06-29; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Ocular Injury; Blast Injuries
MeSH Terms: conditions — Eye Injuries; Blast Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: fireworks eye injury — patients presented with eye injury during festivals due to fireworks

SUMMARY:
The aim of this study is to explore and report the epidemiology and outcome of fireworks ocular injuries in Upper Egypt.

Primary outcome : type and severity of injury of fireworks eye trauma during festives.

Secondary outcome: demography, complications, and final visual outcome of fireworks eye injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending ocular emergency unit with fireworks eye injury during different festivals in 2024

Exclusion Criteria:

* patients presented with non-fireworks ocular injuries

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients attending ocular emergency unit with eye injury during different festivals in 2024
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
epidemiology and outcome of fireworks eye injury | through study completion, an average of 1 year
  Age, gender, laterality, type of eye injury, complications, final visual outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided